CLINICAL TRIAL: NCT05724160
Title: Using Non-Weightbearing Stationary Elliptical Machines and Virtual Reality for Patients with Chronic Nonspecific Low Back Pain; a Prospective Clinical Trial
Brief Title: Using Non-Weightbearing Stationary Elliptical Machines for Patients with Chronic Low Back Pain
Acronym: Cubii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fitness Cubed Inc. (Unknown)
Responsible Party: Principal Investigator, Soheil Ashkani Esfahani, Director, Foot and Ankle Research and Innovation Laboratory, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022P001905
Record Dates: First submitted 2023-01-12; First posted 2023-02-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Chronic Low-back Pain; Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 32 patients with non-specific low back pain will be allocated to the physiotherapy group.
  32 patients with non-specific low back pain will be allocated to the physiotherapy + sitting elliptical group. They will be receive routine physiotherapy care based on the protocols for non-specific low back pain and using the ellipticals will not affect the process of the treatment.
Masking Description: No groups will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSLBP treated with Physiotherapy (Other): 32 patients with non-specific low back pain receiving routine protocol-based physiotherapy care by an expert.
  Interventions: Other: Physiotherapy Protocol
- NSLBP treated with Physiotherapy + Sitting ellipticals (Other): 32 patients with non-specific low back pain receiving routine protocol-based physiotherapy care by an expert together with planned training using sitting ellipticals
  Interventions: Other: Using sitting ellipticals; Other: Physiotherapy Protocol

INTERVENTIONS:
Other: Using sitting ellipticals — Patients will receive routine physiotherapy protocols as well as Non-weightbearing stationary elliptical
  Other Names: Cubii Ellipticals
  Arms: NSLBP treated with Physiotherapy + Sitting ellipticals
Other: Physiotherapy Protocol — Routine physiotherapy protocol
  Other Names: Physiotherapy

SUMMARY:
The goal of this clinical trial is to assess the effect of non-weightbearing stationary ellipticals (Cubii, Fitness Cubed, Inc.) on patient well-being with chronic lower back pain (CLBP). The main questions it aims to answer are:

1. Assess the effect of non-weightbearing stationary ellipticals on clinical outcomes inclduing vital signs, pain, disability, analgesic use, mental health, abdominal muscle strength, and compliance in patients with CLBP.
2. Assess the effect of placing the patients into an interactive virtual environment during the exercise sessions on the outcomes of the program

Participants will participate in 60 minute training sessions to see if there are effects to their CLBP.

DETAILED DESCRIPTION:
There are controversies on whether exercise is more effective than placebo among different clinical studies specifically in acute LBP; however, in CLBP cases, evidence strongly recommends that exercise is more effective than conservative treatment on pain and functional abilities, especially individually designed exercise programs for stabilizing and strengthening. The aims of the present study are:

1. to assess the effect of non-weightbearing stationary ellipticals (Cubii, Fitness Cubed Inc.) on clinical outcomes including vital signs, pain, disability, analgesic use, mental health, abdominal muscle strength, and compliance in patients with CLBP
2. to assess the effect of placing the patients into an interactive virtual environment during the exercise sessions on the outcomes of the program.

The training sessions will be up to 60 minutes and will include a) introduction to the goals of the session (5 minutes), b) warm-up and stretching (10 minutes), c) low resistance flat road cycling (low resistance, low cadence; 10 minutes), d) flat road cycling (high resistance, low cadence; 10 minutes), e) flat road sprint (low resistance, high cadence; 10 minutes), f) warm-down, whole-body stretching, questions and answers (Q&A; 10-15 minutes) obtained from investigations on the similar topic. The training sessions will be supervised by both an expert clinical researcher with MD degree who is familiar with healthcare principles for these patients and also by a US licensed board-certified orthopaedic surgeon, who is responsible for providing routine orthopaedic care for the patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years and CLBP (>12 wk) located between the costal margins and inferior gluteal folds.

Exclusion Criteria:

* The presence of a postural abnormality contributing to the diagnosis reported by an expert spine surgeon
* Pain radiating below the knee, past medical history or current symptomatic lumbar disc hernia or fracture based on expert reports (i.e. orthopedic surgeon or radiologist)
* History of back surgery, inflammatory joint disease, severe osteoporosis
* A metabolic disease affecting the CLBP, or neuromuscular disease (as assessed by the American College of Sports Medicine pre-exercise screening tool for cardiovascular risk factors prior to entry into an exercise program)
* Pregnancy
* Ankle and foot injuries inhibiting them from cycling recently (<3 mo.)
* Participation in another exercise program or physiotherapy (i.e., manipulation, mobilization, range of motion, massage).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Heart rate | 8 weeks
  Heart rate in beats/minute
Pain Visual Analogue Scale (VAS) | 8 weeks
  Pain scores based on the Visual Analogue Scale 0-10
Pain Catastrophizing Scale (PCS) | 8 weeks
  Mental health based on the Pain Catastrophizing Scale (PCS). 13-item questionnaire to identify catastrophic thoughts or feelings in relation to painful experiences. The total score ranges from 0 to 52, with high scores indicating that more catastrophic thoughts or feelings are experienced.
Oswestry Low Back Pain Disability Index (ODI) | 8 weeks
  Measure of disability based on the Oswestry Low Back Pain Disability Index (ODI). Version 2, 10-item questionnaire on how LBP affects aspects of their life (0%-100% scoring.
Transversus abdominis endurance (TAE) | 8 weeks
  Abdominal strength based on Transversus abdominis endurance (TAE). Holding or tonic capacity of transversus abdominis measured by the number of 10-second holds (up to 10) using pressure biofeedback in prone position.
Fear-Avoidance Beliefs Questionnaire (FABQ) | 8 weeks
  Patient's beliefs about the potential harm of work or general physical activity to their back pain. Two subscales within the FABQ have been identified, a 7-item work subscale score (FABQw, score range 0-42), and a 4-item physical activity subscale score (FABQa, score range 0-24)
Patient reported outcome measures (PROM) | 8 weeks
  PROMIS-29 profile v1.0 (for Physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with social role, pain inference (+pain inference short form 6b), pain intensity, depression, mood and anxiety.

SECONDARY OUTCOMES:
Duration of exercise in each session | 8 weeks
  Duration of exercise in each session as feedback on the session
Satisfaction rate (0-10) | 8 weeks
  Satisfaction rate (0-10) as feedback on the session
Compliance (duration of continuing the sessions) | 8 weeks
  Compliance (duration of continuing the sessions) as feedback on the session
Intention to continue the sessions (0-10) | 8 weeks
  Intention to continue the sessions (0-10) as feedback on the session
Distance passed on the stationary elliptical | 8 weeks
  Distance passed on the stationary elliptical as elliptical measurement in kilometers
Total strides | 8 weeks
  Total strides as elliptical measurement
Time series of the stride/minute | 8 weeks
  Time series of the stride/minute as elliptical measurement
Average strides/minute | 8 weeks
  Average strides/minute as elliptical measurement
Distance traveled in each section | 8 weeks
  Distance traveled in each section as elliptical measurement in kilometers

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All data acquired as specified by this protocol will be maintained and monitored by approved study staff. Approved study staff will be responsible for collecting the signed consent forms. All electronic data and subject information will be secured on non-networking password protected computers; all paperwork will be secured in locked filing cabinets. All electronic data and subject information will be secured in REDCap and will be secured on non-networking password protected computers to which only study staff will have access; all paper work will be secured in locked filing cabinets.

REFERENCES:
- [Background] Andersson GB. Epidemiological features of chronic low-back pain. Lancet. 1999 Aug 14;354(9178):581-5. doi: 10.1016/S0140-6736(99)01312-4. PMID 10470716
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Patrick N, Emanski E, Knaub MA. Acute and chronic low back pain. Med Clin North Am. 2014 Jul;98(4):777-89, xii. doi: 10.1016/j.mcna.2014.03.005. PMID 24994051
- [Background] Henchoz Y, Kai-Lik So A. Exercise and nonspecific low back pain: a literature review. Joint Bone Spine. 2008 Oct;75(5):533-9. doi: 10.1016/j.jbspin.2008.03.003. Epub 2008 Sep 17. PMID 18801686
- [Background] Illes ST. [Low back pain: when and what to do]. Orv Hetil. 2015 Aug 16;156(33):1315-20. doi: 10.1556/650.2015.30232. Hungarian. PMID 26256495
- [Background] Hayden JA, van Tulder MW, Malmivaara AV, Koes BW. Meta-analysis: exercise therapy for nonspecific low back pain. Ann Intern Med. 2005 May 3;142(9):765-75. doi: 10.7326/0003-4819-142-9-200505030-00013. PMID 15867409
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] Marshall PW, Kennedy S, Brooks C, Lonsdale C. Pilates exercise or stationary cycling for chronic nonspecific low back pain: does it matter? a randomized controlled trial with 6-month follow-up. Spine (Phila Pa 1976). 2013 Jul 1;38(15):E952-9. doi: 10.1097/BRS.0b013e318297c1e5. PMID 23615384
- [Background] Chulliyil SC, Sheth MS, Vyas NJ. EFFECT OF TREADMILL WALKING VERSUS STATIONARY CYCLING ON PAIN, TRANSVERSUS ABDOMINIS ENDURANCE, DISABILITY & QUALITY OF LIFE IN NON-SPECIFIC CHRONIC LOW BACK PAIN: A QUASI EXPERIMENTAL STUDY. Int J Physiother Res. 2018;6(5):2848-56.
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Kisner C, Colby L. The spine: exercise interventions. Therapeutic exercise: foundations and techniques 5th ed Philadelphia: FA Davis Company. 2007:439-81.